CLINICAL TRIAL: NCT07075718
Title: Phase 2/Phase 3 Trial to Evaluate the Safety and Efficacy of the Second Generation Travoprost Intracameral Implant
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: GLK-102-01
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Glaucoma
Keywords: open-angle glaucoma; ocular hypertension
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Period 1 (Cohort A) (Experimental): Single-arm, open-label portion of Phase 2; subjects will receive second generation travoprost intracameral implant (plus placebo eyedrops BID) in the study eye and be followed for 36 months
  Interventions: Drug: Gen 2 Travoprost Intracameral Implant
- Period 2 (Cohort B) Gen 2 Travoprost Intracameral Implant Arm (Experimental): Randomized, double-masked, active-controlled Phase 2 portion of the trial; subjects will receive second generation travoprost intracameral implant (plus placebo eyedrops BID) in the study eye and be followed for 36 months
  Interventions: Drug: Gen 2 Travoprost Intracameral Implant; Other: Placebo eye drops
- Period 2 (Cohort B) Timolol Arm (Active Comparator): Randomized, double-masked, active-controlled, Phase 2 portion of the trial; subjects will administer timolol 0.5% eye drops BID (plus sham procedure) in the study eye and be followed for 36 months
  Interventions: Drug: Timolol eye drops 0.5%; Procedure: Sham Procedure
- Period 3 (Cohort X) Gen 2 Travoprost Intracameral Implant Arm (Experimental): Randomized, double-masked, active-controlled, Phase 3 portion of the trial; subjects will receive second generation travoprost intracameral implant (plus placebo eyedrops BID) in the study eye and undergo an exchange procedure at month 12 and be followed for an additional 12 months
  Interventions: Drug: Gen 2 Travoprost Intracameral Implant; Other: Placebo eye drops
- Period 3 (Cohort X) Timolol Arm (Active Comparator): Randomized, double-masked, active-controlled, Phase 3 portion of the trial; subjects will administer timolol 0.5% eye drops BID (plus sham procedure) in the study eye and undergo a sham exchange procedure at month 12 and be followed for an additional 12 months
  Interventions: Drug: Timolol eye drops 0.5%; Procedure: Sham Procedure
- Period 3 (Cohort Y) Gen 2 Travoprost Intracameral Implant Arm (Active Comparator): Randomized, double-masked, active-controlled, Phase 3 portion of the trial, subjects will receive second generation travoprost intracameral implant (plus placebo eyedrops BID) in the study eye and undergo an exchange procedure at month 24 and be followed for an additional 12 months
  Interventions: Drug: Gen 2 Travoprost Intracameral Implant; Other: Placebo eye drops
- Period 3 (Cohort Y) Timolol Arm (Active Comparator): Randomized, double-masked, active-controlled, Phase 3 portion of the trial; subjects will receive timolol 0.5% eye drops BID (plus sham procedure) in the study eye and undergo a sham exchange procedure at month 24 and be followed for an additional 12 months
  Interventions: Drug: Timolol eye drops 0.5%; Procedure: Sham Procedure
- Period 3 (Cohort Z) Gen 2 Travoprost Intracameral Implant Arm (Experimental): Randomized, double-masked, active-controlled, Phase 3 portion of the trial, subjects will receive second generation travoprost intracameral implant (plus placebo eyedrops BID) in the study eye and undergo an exchange procedure at month 36 and be followed for an additional 12 months
  Interventions: Drug: Gen 2 Travoprost Intracameral Implant
- Period 3 (Cohort Z) Timolol Arm (Active Comparator): Randomized, double-masked, active-controlled, Phase 3 portion of the trial; subjects will administer timolol 0.5% eye drops BID (plus sham procedure) in the study eye and undergo an sham exchange procedure at month 36 and be followed for an additional 12 months
  Interventions: Drug: Timolol eye drops 0.5%; Other: Placebo eye drops

INTERVENTIONS:
Drug: Gen 2 Travoprost Intracameral Implant — travoprost
  Other Names: Gen 2 Travoprost Intraocular Implant
  Arms: Period 1 (Cohort A); Period 2 (Cohort B) Gen 2 Travoprost Intracameral Implant Arm; Period 3 (Cohort X) Gen 2 Travoprost Intracameral Implant Arm; Period 3 (Cohort Y) Gen 2 Travoprost Intracameral Implant Arm; Period 3 (Cohort Z) Gen 2 Travoprost Intracameral Implant Arm
Drug: Timolol eye drops 0.5% — timolol 0.5%
  Other Names: Timolol maleate ophthalmic solution, 0.5%
  Arms: Period 2 (Cohort B) Timolol Arm; Period 3 (Cohort X) Timolol Arm; Period 3 (Cohort Y) Timolol Arm; Period 3 (Cohort Z) Timolol Arm
Procedure: Sham Procedure — sham implant administration
  Arms: Period 2 (Cohort B) Timolol Arm; Period 3 (Cohort X) Timolol Arm; Period 3 (Cohort Y) Timolol Arm
Other: Placebo eye drops — artificial tears
  Arms: Period 2 (Cohort B) Gen 2 Travoprost Intracameral Implant Arm; Period 3 (Cohort X) Gen 2 Travoprost Intracameral Implant Arm; Period 3 (Cohort Y) Gen 2 Travoprost Intracameral Implant Arm; Period 3 (Cohort Z) Timolol Arm

SUMMARY:
Evaluate the Safety and Efficacy of the Second Generation Travoprost Intracameral Implant

DETAILED DESCRIPTION:
Evaluate the Safety and Efficacy of the Second Generation Travoprost Intracameral Implant Compared to Timolol Ophthalmic Solution 0.5% Administered Twice Daily in Subjects with Open-Angle Glaucoma or Ocular Hypertension

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of open-angle glaucoma or ocular hypertension in the study eye

Exclusion Criteria:

* Prior incisional glaucoma surgery in the study eye
* Prior argon laser trabeculoplasty (ALT) in the study eye
* Prior minimally invasive glaucoma (MIGS) surgery in the study eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2032-03 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure (IOP) | 3 months
  Change from baseline in diurnal IOP in the study eye at 8AM and 10AM at each of Day 11, Week 6, and Month 3 visits

CONTACTS AND LOCATIONS:
Overall Officials: Luis G. Vargas, MD, Study Chair — Glaukos Corporation
Locations (3):
- United States (3):
  - Glaukos Investigative Site, Grand Junction, Colorado
  - Glaukos Investigative Site, Oklahoma City, Oklahoma
  - Glaukos Clinical Site, El Paso, Texas

IPD SHARING:
Plan to Share IPD: No